CLINICAL TRIAL: NCT02781571
Title: A Phase 2, Multicenter, Open-Label Study to Evaluate the Efficacy and Safety of Sofosbuvir/Velpatasvir Fixed Dose Combination in Subjects With Chronic HCV Infection Who Have Received a Liver Transplant
Brief Title: Sofosbuvir/Velpatasvir Fixed Dose Combination in Participants With Chronic Hepatitis C Virus Infection Who Have Received a Liver Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-342-2104; 2016-000416-15 (EudraCT Number)
Record Dates: First submitted 2016-05-20; First posted 2016-05-24 (Estimated); Results first posted 2018-08-21 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-07

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- SOF/VEL (Experimental): SOF/VEL FDC for 12 weeks
  Interventions: Drug: SOF/VEL

INTERVENTIONS:
Drug: SOF/VEL — 400/100 mg tablet administered orally once daily
  Other Names: Epclusa®; GS-7977/GS-5816

SUMMARY:
The primary objectives of this study are to evaluate the efficacy, safety, and tolerability of sofosbuvir /velpatasvir (SOF/VEL) fixed-dose combination (FDC) in participants with chronic hepatitis C virus (HCV) who have received a liver transplant.

ELIGIBILITY:
Key Inclusion Criteria:

* History of chronic HCV infection (≥ 6 months)
* HCV genotype 1, 2, 3, 4, 5, 6, or indeterminate
* Liver transplant ≥ 3 months prior to screening
* Male and nonpregnant/ non-lactating female individuals without cirrhosis or with compensated cirrhosis

Key Exclusion Criteria:

* History of clinically significant illness or any other medical disorder that may interfere with individual's treatment, assessment or compliance with the protocol,
* Co-infection with HIV or hepatitis B virus
* Known hypersensitivity to study medication,
* Use of any prohibited concomitant medications as within with window before the Day 1 visit.
* De novo or recurrent hepatocellular carcinoma posttransplant

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2016-07-27 (Actual); Primary Completion 2017-07-28 (Actual); Study Completion 2017-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (15):
- Spain (8):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Reina Sofía University Hospital, Córdoba
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Ramón Y Cajal, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
  - La Fe Hospital, Valencia
  - Hospital Clinico Zaragoza, Zaragoza
- Switzerland (2):
  - Universität Bern, Bern
  - University Hospital Zurich, Zurich
- United Kingdom (5):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Royal Infirmary of Edinburgh, Edinburgh
  - St James University Hospital, Leeds
  - Kings College Hospital, London
  - Royal Free Hampstead NHS Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Background] Agarwal K, Castells L, Mullhaupt B, Rosenberg WMC, McNabb B, Arterburn S, Camus G, McNally J, Stamm LM, Brainard DM, Mani Subramanian G, Marino Z, Dufour JF, Forns X. Sofosbuvir/velpatasvir for 12 weeks in genotype 1-4 HCV-infected liver transplant recipients. J Hepatol. 2018 Sep;69(3):603-607. doi: 10.1016/j.jhep.2018.05.039. Epub 2018 Jun 8. PMID 29886154

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Spain, Switzerland, and the United Kingdom. The first participant was screened on 27 July 2016. The last study visit occurred on 28 July 2017.
Pre-assignment Details: 85 participants were screened.
Groups:
- SOF/VEL: Sofosbuvir/Velpatasvir (SOF/VEL) (400/100 mg) fixed-dose combination (FDC) tablet orally once daily for 12 weeks in participants with chronic HCV infection who received a liver transplant
Period: Overall Study
Arm/Group | SOF/VEL
Started | 79
Completed | 79
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who took at least 1 dose of the study drug.
Groups:
- SOF/VEL: SOF/VEL (400/100 mg) FDC tablet orally once daily for 12 weeks in participants with chronic HCV infection who received a liver transplant
Arm/Group | SOF/VEL
Number analyzed (Participants) | 79
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 77
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 65
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 41
  Switzerland | 7
  Spain | 31
IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 39
    CT | 34
    TT | 6
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.4 (0.55)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 18
  ≥ 800,000 IU/mL | 61
HCV genotype [Count of Participants; unit: Participants]
  Genotype 1 | 37
  Genotype 2 | 3
  Genotype 3 | 35
  Genotype 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Cessation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: all enrolled participants who took at least 1 dose of the study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 79
percentage of participants | 96.2 [89.3 to 99.2]

2. Primary Outcome: Percentage of Participants Who Prematurely Discontinued Study Drug Due to Any Adverse Event
Time Frame: Up to 12 weeks
Population: Safety Analysis Set: participants who took at least 1 dose if the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 79
percentage of participants | 1.3

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 4 Weeks After Cessation of Therapy (SVR4)
Description: SVR4 was defined as HCV RNA < LLOQ at 4 weeks after stopping study treatment.
Time Frame: Posttreatment Week 4
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 79
Percentage of participants | 97.5 [91.2 to 99.7]

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 2
Time Frame: Week 2
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 79
percentage of participants | 40.5 [29.6 to 52.1]

5. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 4
Time Frame: Week 4
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 78
percentage of participants | 85.9 [76.2 to 92.7]

6. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 8
Time Frame: Week 8
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 78
percentage of participants | 98.7 [93.1 to 100.0]

7. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 12
Time Frame: Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 78
percentage of participants | 100.0 [95.4 to 100.0]

8. Secondary Outcome: HCV RNA at Week 2
Time Frame: Week 2
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL
Number analyzed (Participants) | 75
log10 IU/mL | 1.59 (0.596)

9. Secondary Outcome: HCV RNA at Week 4
Time Frame: Week 4
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL
Number analyzed (Participants) | 78
log10 IU/mL | 1.23 (0.251)

10. Secondary Outcome: HCV RNA at Week 8
Time Frame: Week 8
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL
Number analyzed (Participants) | 77
log10 IU/mL | 1.15 (0.00)

11. Secondary Outcome: HCV RNA at Week 12
Time Frame: Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL
Number analyzed (Participants) | 78
log10 IU/mL | 1.15 (0.00)

12. Secondary Outcome: Change From Baseline in HCV RNA at Week 2
Time Frame: Baseline; Week 2
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL
Number analyzed (Participants) | 75
log10 IU/mL | -4.75 (0.635)

13. Secondary Outcome: Change From Baseline in HCV RNA at Week 4
Time Frame: Baseline; Week 4
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL
Number analyzed (Participants) | 78
log10 IU/mL | -5.13 (0.551)

14. Secondary Outcome: Change From Baseline in HCV RNA at Week 8
Time Frame: Baseline; Week 8
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL
Number analyzed (Participants) | 77
log10 IU/mL | -5.20 (0.548)

15. Secondary Outcome: Change From Baseline in HCV RNA at Week 12
Time Frame: Baseline; Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL
Number analyzed (Participants) | 78
log10 IU/mL | -5.22 (0.554)

16. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as
  On-treatment virologic failure:
  * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ on 2 consecutive measurements while on treatment), or
  * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
  * Non-response (HCV RNA persistently ≥ LLOQ through 12 weeks of treatment)
  Virologic relapse:
  * HCV RNA ≥ LLOQ during the post-treatment period having achieved HCV RNA < LLOQ at end of treatment, confirmed with 2 consecutive values or last available post-treatment measurement
Time Frame: Up to Posttreatment Week 12
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 79
percentage of participants | 2.5

ADVERSE EVENTS:
Time Frame: Up to 12 weeks plus 30 days
Description: Safety Analysis Set: participants who took at least 1 dose of the study drug.
Arm/Group | SOF/VEL
All-Cause Mortality (participants affected / at risk) | 0/79
Serious Adverse Events (participants affected / at risk) | 3/79
Other Adverse Events (participants affected / at risk) | 42/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL (N=79)
Pneumonia klebsiella (Infections and infestations) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL (N=79)
Diarrhoea (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 6
Asthenia (General disorders) | 5
Fatigue (General disorders) | 16
Influenza (Infections and infestations) | 5
Viral upper respiratory tract infection (Infections and infestations) | 5
Decreased appetite (Metabolism and nutrition disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Headache (Nervous system disorders) | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2016-02-19): https://cdn.clinicaltrials.gov/large-docs/71/NCT02781571/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT02781571/SAP_001.pdf